CLINICAL TRIAL: NCT00264992
Title: The Cytokine Paired Footprint of Successful Implantation
Brief Title: Implantation and Cytokine Expression
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Other Study IDs: ICE-STUDY
Record Dates: First submitted 2005-12-09; First posted 2005-12-13 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Infertility
Keywords: embryo implantation, in vitro fertilization,; cytokine expression
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Implantation failure of the embryo might be the result from the environment in the uterus. Proteins (cytokines) are screted by the endometrium which can result in a pro or anti inflammatory environment. The aim of this study is to identify pre-implantation endometrial and embryo cytokine expression profiles associated with successful and unsuccessful embryo implantation in assisted reproduction cycles.

DETAILED DESCRIPTION:
Rationale:

Failure of the transferred embryo to implant remains the most important limiting factor determining IVF success rates. It is hypothesed that implantation failure following IVF treatment may be caused by abnormal cytokine expression by embryos and endometrium and by subclinical bacterial vaginosis. Analysis of cytokine expression in the culture media of embryos and in the endometrium during 'the window of implantation' offers the opportunity to study the cross-talk between the embryo and endometrium and identify optimal cytokine expression patterns. Increased knowledge of cytokine interaction and the impact of bacterial vaginosis on cytokine expression may serve as the basis from which to develop and apply treatment regimens to improve embryo selection and endometrial preparation.

Objective:

The aim of this study is to identify pre-implantation endometrial and embryo cytokine expression profiles associated with successful and unsuccessful implantation.

Study design:

The study design is a prospective, mono-center, observational cohort study. Study population: We will aim to include at least 160 women initiating their first or second IVF/ ICSI cycle. A subgroup of forty women will be invited for endometrial secretion aspiration in a natural cycle as well.

Main study parameters/endpoints:

For research purposes, transcervical aspiration of endometrial secretion will be performed. An endocervical swab will be taken to assess the existence of bacterial vaginosis. A single ultrasound measurement of uterine artery pulsatile resistance will be made (by pulsed Doppler) and endometrium thickness will be measured. The embryo transfer and IVF/ ICSI treatment will be performed as usual. The main study parameter is the cytokine profile in the endometrium and from the embryo culture medium, measured with Luminex (a multiplex immunoassay). Implantation rate, ultrasound measurements and bacterial vaginosis will be correlated to the cytokine profile. The cytokine profile from the endometrium will be compared with the cytokine profile from the supernatant of the embryo. In a reference group the cytokine profile in the endometrial secretion in a natural cycle will be compared to the cytokine profile in a IVF/ ICSI treatment cycle.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The theoretical risk associated with this study might be disruption of embryo implantation. However, our group has developed a technique of obtaining endometrial material at the time of embryo transfer which, as we have previously shown, does not disrupt the process of implantation. The burden is minimal; patients will not have to make an extra visit to the hospital. The investigations are painless and will not take more than a few minutes. No side effects or risks have been reported.

ELIGIBILITY:
Inclusion Criteria:

* all women starting their first or second IVF/ ICSI treatment cycle.

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Macklon, Prof. dr., Principal Investigator — UMC Utrecht
Locations (1):
- University Medical center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] van der Gaast MH, Beier-Hellwig K, Fauser BC, Beier HM, Macklon NS. Endometrial secretion aspiration prior to embryo transfer does not reduce implantation rates. Reprod Biomed Online. 2003 Jul-Aug;7(1):105-9. doi: 10.1016/s1472-6483(10)61737-3. PMID 12930588
- [Derived] Boomsma CM, Kavelaars A, Eijkemans MJ, Lentjes EG, Fauser BC, Heijnen CJ, Macklon NS. Endometrial secretion analysis identifies a cytokine profile predictive of pregnancy in IVF. Hum Reprod. 2009 Jun;24(6):1427-35. doi: 10.1093/humrep/dep011. Epub 2009 Feb 19. PMID 19228761